CLINICAL TRIAL: NCT04627064
Title: A Phase I/IB Trial of Abemaciclib Alone or in Combination With MK-6482 in Advanced Renal Cell Carcinoma
Brief Title: ABEMA Alone or in COMBO With MK-6482
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Toni Choueiri, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-284; 5P50CA101942-20 (NIH)
Record Dates: First submitted 2020-10-09; First posted 2020-11-13 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — abemaciclib; belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib-Arm 1 (Experimental): Arm 1
  * Abemaciclib will be taken at a standard recommended starting dose 2X daily during 28 day study cycles and will be taken until radiographic progression, unacceptable toxicity or withdrawal.
  * Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks, in both Arm 1 and Arm 2.
  Interventions: Drug: Abemaciclib
- Abemaciclib and MK-6482-Arm 2 (Experimental): Arm 2
  * Arm 2 will start enrolling only after there is experience with Arm 1 to see what abemaciclib effects are when given alone,
  * Dose escalation will occur following a 3+3 design.
  * Abemaciclib will be taken 2X daily uring 28 day study cycle
  * MK-6482 will be taken 1x daily during 28 day study cycle
  * Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks, in both arms.
  Interventions: Drug: Abemaciclib; Drug: MK-6482

INTERVENTIONS:
Drug: Abemaciclib — Tablet taken orally
  Other Names: Verzenio
Drug: MK-6482 — Tablet taken orally
  Other Names: HIF-2α inhibitor
  Arms: Abemaciclib and MK-6482-Arm 2

SUMMARY:
This research study will assess whether abemaciclib alone or in combination with MK-6482 are safe and effective in slowing down the growth of clear cell renal cell carcinoma (ccRCC).

The names of the study drugs in this investigational combination are:

* Abemaciclib
* MK-6482

DETAILED DESCRIPTION:
This a two-arm, non-randomized phase 1/1B trial aiming at assessing the safety and activity of abemaciclib alone (arm 1), and abemaciclib plus MK-6482 (arm 2) in patients with advanced refractory clear-cell renal cell carcinoma (croc).

A Phase I clinical trial tests the safety of an investigational drug or drug combination and also tries to define the appropriate dose of the investigational drug or drug combination to use for further studies. "Investigational" means that the drug is being studied.The U.S. Food and Drug Administration (FDA) has not approved either abemaciclib or MK-6482 for renal (kidney) cancer but abemaciclib has been approved to treat other forms of cancer.

Abemaciclib is in a class of drugs known as CDK4 & 6 inhibitors. These proteins control how fast cells grow and divide and are found on both normal and cancer cells. They become overactive in cancer cells causing cells to grow and divide uncontrollably. Abemaciclib blocks these proteins just as the cells start to grow and divide and in other cancers has been shown to slow down cancer cell growth and division, causing cancer cells to become inactive or even die.

MK-6482 is an oral, first-in-class selective small-molecule inhibitor that targets hypoxia-inducible factor (HIF)-2a, which promotes the growth of new vessels that fuel kidney cancer.

This study is looking at two different treatments:

* Arm 1 - abemaciclib alone:

  * To determine the response rate of abemaciclib alone in patients with advanced ccRCC
* Arm 2 - combination therapy of abemaciclib and MK-6482

  * To determine the maximum dose of abemaciclib and MK-6482 in combination.
  * To determine the response rate of abemaciclib and MK-6482 in patients with advanced ccRCC.

The research study procedures include screening for eligibility, study treatment, participant evaluations and safety follow-up visits, in addition to general health status follow-up after study treatment. It is estimated that participants will receive 12 to 18 months of study treatment and 3 months of safety follow-up, totaling about 15 to 21 months from the start of study treatment. After the safety follow-up visits, the study doctor may request that participants return to clinic for additional tumor assessments or his/her staff will contact participants about every 6 months to follow their health status and find out about any anticancer treatments participants may have begun after study treatment.

It is expected that about 40 people will take part in this research study.

The pharmaceutical company Eli Lilly is supporting this research study by providing funding for the research study, tests required for research purposes only, and the study drugs. The pharmaceutical company Merck is supporting this research study by providing study drug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable advanced or metastatic renal cell carcinoma with clear cell component. Patients with extensive sarcomatoid histology are accepted.
* Participants must have failed or developed an intolerance to at least 1 prior anti-VEGFR systemic therapy and 1 immune checkpoint inhibitor for metastatic RCC. No limit on the number of prior lines of therapies.
* Measurable disease as per RECIST 1.1. See section 12 for the evaluation of measurable disease.
* Age ≥ 18 years
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must undergo fresh tumor biopsy unless medically unsafe or not feasible.
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥10g/dL (transfusions allowed)

    * Total bilirubin ≤2.0 x institutional upper limit of normal with the following exception: patients with known Gilbert disease should have a serum bilirubin ≤ 3 x ULN
    * AST(SGOT)/ALT(SGPT)≤3.0 × institutional upper limit of normal with the following exception: patients with known liver metastases should have AST and ALT

      ≤ 5 x ULN
    * Creatinine clearance ≥30 mL/min/1.73 m2 according to the Cockcroft-Gault equation. (APPENDIX F)
    * Urine protein/creatinine ratio (UPC ratio) ≤2
* Women of child-bearing potential and men must agree to use adequate contraception (intrauterine device or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and 6 months after completion abemaciclib plus MK- 6482 and at least 3 weeks after the completion of abemaciclib administration. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection. A negative pregnancy serum test should be obtained within 7 days of therapy initiation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation.. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion abemaciclib plus MK-6482 and at least 3 weeks after the completion of abemaciclib administration.
* Ability to swallow oral medications
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

A patient will be excluded from the study if he or she meets any of the following criteria:

* Patients receiving any other investigational agents.
* Patients who received prior CDK4/6 inhibitors.
* For Arm 2 only, patients who have received prior HIF-2α inhibitor.
* Participants who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 4 effective half-lives prior to starting study drug or who have not recovered from side effects of such therapy to grade 1 or less (except for non-clinically significant laboratory abnormalities).
* Patients must have discontinued all biologic therapy including therapeutic antibodies at least 28 days before C1D1.
* Participants who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy to at least grade 1.
* O2 saturation <92% by arterial blood gas analysis or pulse oximetry on room air
* Untreated deep vein thrombosis or pulmonary embolism, or event of deep vein thrombosis or pulmonary embolism within 2 weeks of treatment start. Patient should be on at least 1 week of anticoagulation before C1D1.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea)."
* Patient with active systemic bacterial infection (requiring IV antibiotics at the time of initiating study treatment), fungal infection, or detectable viral infection. Patients with known viral infection (such as HIV) are excluded given the potential for interactions between antiretroviral agents and abemaciclib, and the potential for increased risk of lifethreatening infection with therapy that is myelosuppressive. If you are not known to have HIV, a HIV test is required.
* Patients with known Hepatitis B or Hepatitis C infection are excluded only if there is evidence of active infection (detectable Hepatitis B surface antigen, detectable Hepatitis C RNA).
* Prior allogenic stem cell or solid organ transplant.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Participants who have undergone major surgery ≤ 4 weeks (28 days) prior to starting study drug(s) or who have not recovered from side effects of such therapy.
* Participants who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
* Other malignancy diagnosed within 2 years of first study treatment unless negligible risk of metastases or death according to the investigator (included but not limited to carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma, or other malignancy not deemed to impact patients 5-year life expectancy).
* Has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), sudden cardiac arrest.
* Has had any major cardiovascular event within 6 months prior to study drug administration iincluding but not limited to: myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic event or New York Heart Association Class III or IV heart failure. Patients with history of DVT or PE are eligible provided DVT or PE occurred at least 2 weeks prior to C1D1 and anticoagulation has been initiated at least 1 week before C1D1.
* History of symptomatic respiratory condition considered clinically significant by the investigator. History of asymptomatic radiation pneumonitis within a previous radiation field is permitted.
* Participants with a known hypersensitivity to the study compounds or to its excipients.
* Participant is unable or unwilling to abide by the study protocol or cooperate fully with the investigator
* Females that are pregnant or lactating
* Participants who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pommelos.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni K Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Meiman D, Skaar TC, Shugg T, Quinney SK. Physiologically Based Pharmacokinetic Model to Assess the Drug-Drug-Gene Interaction Potential of Belzutifan in Combination With Cyclin-Dependent Kinase 4/6 Inhibitors. JCO Precis Oncol. 2025 Jul;9:e2500153. doi: 10.1200/PO-25-00153. Epub 2025 Jul 25. PMID 40712111

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib-Arm 1: Arm 1
  * Abemaciclib will be taken at a standard recommended starting dose 2X daily during 28 day study cycles and will be taken until radiographic progression, unacceptable toxicity or withdrawal.
  * Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks thereafter.
  Abemaciclib: Tablet taken orally
- Abemaciclib and MK-6482-Arm 2: Arm 2
  * Arm 2 will start enrolling only after there is experience with Arm 1 to see what abemaciclib effects are when given alone,
  * Dose escalation will occur following a 3+3 design.
  * Abemaciclib will be taken 2X daily uring 28 day study cycle
  * MK-6482 will be taken 1x daily during 28 day study cycle
  * Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks thereafter.
  Abemaciclib: Tablet taken orally
  MK-6482: Tablet taken orally
Period: Overall Study
Arm/Group | Abemaciclib-Arm 1 | Abemaciclib and MK-6482-Arm 2
Started | 11 | 0 (Arm 2 never opened.)
Completed | 0 | 0 (Arm 2 never opened)
Not Completed | 11 | 0
Not completed — Progressive disease | 8 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Arm1 included 11 patients enrolled on the study and receiving protocol treatment.
  Arm 2 never opened.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abemaciclib-Arm 1 | Abemaciclib and MK-6482-Arm 2 | Total
Number analyzed (Participants) | 11 | 0 | 11
Age, Continuous [Median (Full Range); unit: Years] | 62 [54 to 68] |  | 62 [54 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 7 |  | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 11 |  | 11
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 11 |  | 11
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 |  | 11
Number of Prior Lines of Systemic Therapy [Median (Full Range); unit: number of therapies] | 4 [1 to 9] |  | 4 [1 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Abemaciclib Arm (Arm 1)
Description: ORR is defined as percentage of patients with partial (PR) or complete response (CR) as best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by central review. Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks thereafter.
Time Frame: From the start of protocol treatment until disease progression or deaths. The total duration assessed was up to 3 months, as all patients either progressed, died, or withdrew from the study within that timeframe.
Population: The analysis dataset is comprised of all treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib-Arm 1
Number analyzed (Participants) | 11
Participants | 0

2. Primary Outcome: Objective Response Rate (ORR) in Abemaciclib and MK-6482 Arm (Arm 2)
Description: Percentage of patients with partial (PR) or complete response (CR) as best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by central review. Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks thereafter.
Time Frame: From the start of protocol treatment until disease progression or death
Population: Arm 2 never opened
Arm/Group | Abemaciclib and MK-6482-Arm 2
Number analyzed (Participants) | 0

3. Primary Outcome: Maximum Tolerated Dose (MTD) in Abemaciclib and MK-6482 (Arm 2)
Description: MTD of abemaciclib plus MK-6482, defined as the highest dose studied at which no more than 1 of 6 subjects has experienced a dose limiting toxicity (DLT) in cycle 1.
Time Frame: Cycle 1 of during the combination therapy (Arm 2)
Population: Arm 2 never opened.
Arm/Group | Abemaciclib and MK-6482-Arm 2
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE 5 of Abemaciclib and MK-6482 (Arm 2)
Description: Toxicity will be graded and analyzed using CTCAE version 5. Treatment related AE will define as "Definitely", "Probably" or "Possibly" related to the study drugs.
Time Frame: From start of protocol treatment until 90 days after treatment discontinuation, or until initiation of new cancer-directed treatment, or until death, whichever occurs first.
Population: Arm 2 never opened
Arm/Group | Abemaciclib and MK-6482-Arm 2
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response (DOR) in Patients Who Achieve an Objective Response in Abemaciclib Arm (Arm 1)
Description: The duration of response is defined from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the date of disease progression or death due to any cause. Participants without events reported are censored at the last disease evaluation.
  Response and progression will be evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
  Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks thereafter.
Time Frame: From start of complete response or partial response (whichever is first recorded) until the date of disease progression or death.
Population: No patient achieved an objective response by RECIST 1.1 criteria in Arm 1
Arm/Group | Abemaciclib-Arm 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-free Survival (PFS) in Abemaciclib Arm (Arm 1)
Description: PFS is measured from the start of treatment until documented progression by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) or death from any cause or censored at the last disease evaluation. PFS will be estimated using the method of Kaplan-Meier with 95% confidence intervals.
  Imaging assessments will be performed every 8 weeks during the first six months of the study, then every 12 weeks thereafter.
Time Frame: From trial treatment start to the earlier of progression or death due to any cause. The total duration assessed was up to 3 months, as all patients either progressed, died, or withdrew from the study within that timeframe.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib-Arm 1
Number analyzed (Participants) | 11
months | 1.8 [1.5 to 1.9]

7. Secondary Outcome: Overall Survival (OS) in Abemaciclib Arm (Arm 1)
Description: OS is measured from the start of treatment until date of death from any cause or censored at the date of last follow-up. OS will be estimated using the method of Kaplan-Meier with 95% confidence intervals.
Time Frame: From trial treatment start to death due to any cause or date last known alive, up to 23 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib-Arm 1
Number analyzed (Participants) | 11
months | 9.1 [2.1 to 15.3]

8. Secondary Outcome: Duration of Response (DOR) in Patients Who Achieve an Objective Response in Abemaciclib and MK-6482 Arm (Arm 2)
Description: as for outcome 5
Time Frame: From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the date of disease progression or death due to any cause.
Population: Arm 2 never opened
Arm/Group | Abemaciclib and MK-6482-Arm 2
Number analyzed (Participants) | 0

9. Secondary Outcome: Progression-free Survival (PFS) in Abemaciclib and MK-6482 Arm (Arm 2)
Description: as for outcome 6
Time Frame: From trial treatment start to the earlier of progression or death due to any cause
Population: Arm 2 never opened
Arm/Group | Abemaciclib and MK-6482-Arm 2
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Survival (OS) in Abemaciclib and MK-6482 Arm (Arm 2)
Description: OS is defined the time from the start of treatment until date of death from any cause or censored at the date of last follow-up. OS will be estimated using the method of Kaplan-Meier with 95% confidence intervals.
Time Frame: From trial treatment start to death due to any cause or date last known alive
Population: Arm 2 never opened
Arm/Group | Abemaciclib and MK-6482-Arm 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For "Adverse event" reporting, the time frame was from start of protocol treatment until 90 days after treatment discontinuation, or until initiation of new cancer-directed treatment, or until death (whichever occurred first), up to 3.3 months. For "All-cause mortality" reporting, the time frame was from start of protocol treatment until deaths from any cause or until the date of last follow up for alive patients, up to 23 months.
Description: Adverse events (AE) are graded using Common Terminology Criteria v5.0. Serious AEs include clinically significant AEs that are fatal, life-threatening, hospitalization-requiring, resulting in significant disability/incapacity or congenital anomaly/birth defect or other significant medical events defined by protocol. All other AEs are non-SAEs.
Arm/Group | Abemaciclib-Arm 1
All-Cause Mortality (participants affected / at risk) | 9/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib-Arm 1 (N=11)
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib-Arm 1 (N=11)
Diarrhea (Gastrointestinal disorders) | 9
Creatinine increased (Investigations) | 9
Anemia (Blood and lymphatic system disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Weight loss (Investigations) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Pain (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT04627064/Prot_SAP_000.pdf